CLINICAL TRIAL: NCT02240238
Title: A Phase 1b/2 Dose Escalation and Expansion Trial of NC-6004 (Nanoparticle Cisplatin) Plus Gemcitabine in Patients With Advanced Solid Tumors or Non-Small Cell Lung, Biliary Tract, and Bladder Cancer
Brief Title: Combination Therapy With NC-6004 and Gemcitabine in Advanced Solid Tumors or Non-Small Cell Lung, Biliary and Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NanoCarrier Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NC-6004-004A
Record Dates: First submitted 2014-08-19; First posted 2014-09-15 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — demplatin pegraglumer; Gemcitabine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NC-6004 and Gemcitabine (Experimental)
  Interventions: Drug: NC-6004; Drug: Gemcitabine

INTERVENTIONS:
Drug: NC-6004 — NC-6004 - given at escalating doses of 60, 75, 90, 105, 120, 135, 150, 165, or 180 mg/m2 according to observations of dose-limiting toxicity.
Drug: Gemcitabine — Gemcitabine 1250 mg/m2 will be administered as a 30 minute intravenous infusion on Day 1 after the completion of the NC 6004 infusion and on Day 8 of each cycle.

SUMMARY:
In the dose escalation phase (Part 1), this study will determine the dose-limiting toxicities (DLTs), the maximum tolerated dose (MTD) and recommended Phase 2 (RPII) dose of NC 6004 in combination with gemcitabine.

In the expansion phase of the study (Part 2), study will evaluate the activity, safety, and tolerability at the RPII dose identified in Part 1 in patients with squamous NSCLC, biliary tract, and bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* (Part 1 only) Have a histologically or cytologically confirmed diagnosis of advanced solid tumor that has relapsed or is refractory to standard curative or palliative therapy or has a contraindication to standard therapy.
* (Part 2 only) Cohort 1: Have histologically or cytologically confirmed diagnosis of Stage IV squamous NSCLC and have not received prior chemotherapy or immunotherapy for metastatic disease and are not known to be PD-L1 positive (known high PD-L1 expression defined as Tumor Proportion Score [TPS] greater than or equal to 50%). Patients with known sensitizing mutation in the epidermal growth factor receptor (EGFR) gene or anaplastic lymphoma kinase (ALK) fusion oncogene must have received at least 1 and up to 2 targeted therapies prior to enrollment.
* (Part 2 only) Cohort 2: Have histologically or cytologically confirmed diagnosis of nonresectable, recurrent, or metastatic biliary tract carcinoma (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer, or ampullary carcinoma) and have not received prior systemic anticancer therapy for advanced or metastatic disease.
* (Part 2 only) Cohort 3: Have histologically or cytologically confirmed diagnosis of metastatic or locally advanced TCC of the urinary tract (bladder, urethra, ureter, renal pelvis) (T3b-T4 N0 M0, Tany N1-N3 M0, or Tany Nany M1) and are not candidates for surgery.
* Have measurable disease per RECIST version 1.1.
* Have an ECOG PS of 0 to 1, with the exception of patients in Part 2 (Cohort 3, unfit bladder cancer patients) who may have an ECOG PS of 2
* Adequate bone marrow reserve, liver and renal function
* Have a negative pregnancy test result at Screening for females of childbearing potential
* Male patients must agree to use a condom during treatment and for 90 days after dosing and must agree not to donate sperm for 90 days after dosing
* Women of childbearing potential are willing to agree to use 1 of the study defined effective methods of birth control from the time of study entry to 6 months after the last day of treatment
* Reasonably recovered from preceding major surgery as judged by the investigator or no major surgery within 4 weeks prior to the start of Day 1 treatment

Exclusion Criteria:

* Have received prior platinum therapy in the past 3 months (Part 1) or 6 months in the adjuvant or neoadjuvant setting (Part 2).
* Have received prior cisplatin and gemcitabine concomitantly within the last 6 months or are refractory to cisplatin and gemcitabine.
* Unresolved toxicity from prior radiation, chemotherapy, or other targeted treatment, including investigational treatment
* Have evidence suggesting pulmonary fibrosis or interstitial pneumonia.
* Have a history of thrombocytopenia with complications
* Have known hypersensitivity to platinum compounds or gemcitabine.
* Have uncontrolled diabetes or have hypertension requiring more than 3 medications for control of hypertension.
* Have pre-existing alcoholic liver injury or significant liver disease.
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao da Silva, MD, Principal Investigator
Locations (22):
- United States (10):
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia, Sofia-Grad
  - Complex Oncology Center - Shumen EOOD, Shumen
- Italy (2):
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan
- Poland (2):
  - Wojewodzki Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow
  - Med-Polonia Sp. z o.o., Poznan
- Romania (6):
  - Fundeni Clinical Institute, Bucharest
  - Coltea Clinical Hospital, Bucharest
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncology Center Sfantul Nectarie, Craiova
  - Euroclinic Oncology Center SRL, Iași
  - Institutul Regional de Oncologie Iasi, Iași

REFERENCES:
- [Background] Subbiah V, Grilley-Olson JE, Combest AJ, Sharma N, Tran RH, Bobe I, Osada A, Takahashi K, Balkissoon J, Camp A, Masada A, Reitsma DJ, Bazhenova LA. Phase Ib/II Trial of NC-6004 (Nanoparticle Cisplatin) Plus Gemcitabine in Patients with Advanced Solid Tumors. Clin Cancer Res. 2018 Jan 1;24(1):43-51. doi: 10.1158/1078-0432.CCR-17-1114. Epub 2017 Oct 13. PMID 29030354

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 NC-6004 60 mg/m^2: Participants received intravenous (IV) infusion of NC-6004 60 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 75 mg/m^2: Participants received IV infusion of NC-6004 75 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 90 mg/m^2: Participants received IV infusion of NC-6004 90 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 105 mg/m^2: Participants received IV infusion of NC-6004 105 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 120 mg/m^2: Participants received IV infusion of NC-6004 120 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 135 mg/m^2: Participants received IV infusion of NC-6004 135 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 150 mg/m^2: Participants received IV infusion of NC-6004 150 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 165 mg/m^2: Participants received IV infusion of NC-6004 165 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 1 NC-6004 180 mg/m^2: Participants received IV infusion of NC-6004 180 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles until they experienced disease progression.
- Phase 2 Cohort 1 (NSCLC): Participants with non-small-cell lung cancer (NSCLC) received IV infusion of NC-6004 135 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles for up to 6 cycles.
- Phase 2 Cohort 2 (Biliary Tract Cancer): Participants with biliary tract cancer received IV infusion of NC-6004 135 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles for up to 8 cycles.
- Phase 2 Cohort 3 (Bladder Cancer): Participants with bladder cancer received IV infusion of NC-6004 135 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles for up to 6 cycles.
Period: Phase 1
Arm/Group | Phase 1 NC-6004 60 mg/m^2 | Phase 1 NC-6004 75 mg/m^2 | Phase 1 NC-6004 90 mg/m^2 | Phase 1 NC-6004 105 mg/m^2 | Phase 1 NC-6004 120 mg/m^2 | Phase 1 NC-6004 135 mg/m^2 | Phase 1 NC-6004 150 mg/m^2 | Phase 1 NC-6004 165 mg/m^2 | Phase 1 NC-6004 180 mg/m^2 | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Started | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor termination | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1 NC-6004 60 mg/m^2 | Phase 1 NC-6004 75 mg/m^2 | Phase 1 NC-6004 90 mg/m^2 | Phase 1 NC-6004 105 mg/m^2 | Phase 1 NC-6004 120 mg/m^2 | Phase 1 NC-6004 135 mg/m^2 | Phase 1 NC-6004 150 mg/m^2 | Phase 1 NC-6004 165 mg/m^2 | Phase 1 NC-6004 180 mg/m^2 | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 50 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 14 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 36 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 14 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 11 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — PARTICIPANT WAS DISCONTINUED DUE TO THEIR DETERIORATING CONDITION/CLINICAL PROGRESSION | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — TREATMENT NOT COMPLETED, PARTICIPANT MISSED C6D8 DUE TO PERSONAL REASON | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — PARTICIPANT DECIDED TO TAKE STANDARD OF CARE TREATMENT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — TREATMENT DELAY >14 DAYS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — PARTICIPANT WAS DECLINING CLINICALLY | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — PARTICIPANT DECIDED TO COME OFF THE STUDY AS STUDY WAS ON HOLD. AND DECIDED TO MOVE TO SOC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — CONTINUE WITH ONLY GEMCITABINE, AS PER PARTICIPANT DECISION | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — TREATMENT DELAY GREATER THAN 14 DAYS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 NC-6004 60 mg/m^2 | Phase 1 NC-6004 75 mg/m^2 | Phase 1 NC-6004 90 mg/m^2 | Phase 1 NC-6004 105 mg/m^2 | Phase 1 NC-6004 120 mg/m^2 | Phase 1 NC-6004 135 mg/m^2 | Phase 1 NC-6004 150 mg/m^2 | Phase 1 NC-6004 165 mg/m^2 | Phase 1 NC-6004 180 mg/m^2 | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer) | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 33 | 49 | 12 | 116
Age, Categorical [Count of Participants; unit: Participants] — Population: Three patients in Part 2 were diagnosed incorrectly resulting in assignment to the incorrect cohort. These patients are not included in the cohort summaries.
  Participants
    Phase 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0 | 22
    Phase 1: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1: Between 18 and 65 years | 1 | 0 | 1 | 0 | 1 | 7 | 6 | 1 | 1 | 0 | 0 | 0 | 18
    Phase 1: >=65 years | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 49 | 12 | 94
    Phase 2: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 2: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 32 | 6 | 60
    Phase 2: >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 17 | 6 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Three patients in Part 2 were diagnosed incorrectly resulting in assignment to the incorrect cohort. These patients are not included in the cohort summaries.
  years
    Phase 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0 | 22
    Phase 1 | 54.0 (NA) — One participant | 67.0 (NA) — One participant | 56.0 (NA) — One participant | 69.0 (NA) — One participant | 37.0 (NA) — One participant | 60.0 (7.75) | 33.7 (9.42) | 62.0 (NA) — One participant | 61.0 (NA) — One participant |  |  |  | 52.2 (14.57)
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 49 | 12 | 94
    Phase 2 |  |  |  |  |  |  |  |  |  | 61.7 (9.10) | 62.6 (8.51) | 65.2 (11.87) | 62.6 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Three patients in Part 2 were diagnosed incorrectly resulting in assignment to the incorrect cohort. These patients are not included in the cohort summaries.
  Participants
    Phase 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0 | 22
    Phase 1: Female | 0 | 0 | 1 | 0 | 1 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 11
    Phase 1: Male | 1 | 1 | 0 | 1 | 0 | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 11
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 49 | 12 | 94
    Phase 2: Female |  |  |  |  |  |  |  |  |  | 7 | 18 | 1 | 26
    Phase 2: Male |  |  |  |  |  |  |  |  |  | 26 | 31 | 11 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three patients in Part 2 were diagnosed incorrectly resulting in assignment to the incorrect cohort. These patients are not included in the cohort summaries.
  Participants
    Phase 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0 | 22
    Phase 1: Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 |  |  |  | 4
    Phase 1: Not Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 8 | 3 | 1 | 1 |  |  |  | 15
    Phase 1: Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  | 3
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 49 | 12 | 94
    Phase 2: Hispanic or Latino |  |  |  |  |  |  |  |  |  | 0 | 2 | 0 | 2
    Phase 2: Not Hispanic or Latino |  |  |  |  |  |  |  |  |  | 33 | 47 | 12 | 92
    Phase 2: Unknown or Not Reported |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three patients in Part 2 were diagnosed incorrectly resulting in assignment to the incorrect cohort. These patients are not included in the cohort summaries.
  Participants
    Phase 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0 | 22
    Phase 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
    Phase 1: Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  |  |  | 1
    Phase 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
    Phase 1: Black or African American | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 |  |  |  | 5
    Phase 1: White | 0 | 1 | 1 | 0 | 0 | 7 | 2 | 1 | 1 |  |  |  | 13
    Phase 1: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
    Phase 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 |  |  |  | 3
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 49 | 12 | 94
    Phase 2: American Indian or Alaska Native |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0
    Phase 2: Asian |  |  |  |  |  |  |  |  |  | 0 | 2 | 0 | 2
    Phase 2: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0
    Phase 2: Black or African American |  |  |  |  |  |  |  |  |  | 0 | 1 | 1 | 2
    Phase 2: White |  |  |  |  |  |  |  |  |  | 33 | 44 | 11 | 88
    Phase 2: More than one race |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0
    Phase 2: Unknown or Not Reported |  |  |  |  |  |  |  |  |  | 0 | 2 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] — Population: Three patients in Part 2 were diagnosed incorrectly resulting in assignment to the incorrect cohort. These patients are not included in the cohort summaries.
  cm
    Phase 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0 | 22
    Phase 1 | 187.0 (NA) — One participant | 181.0 (NA) — One participant | 165.10 (NA) — One participant | 189.20 (NA) — One participant | 162.60 (NA) — One participant | 171.08 (12.473) | 175.67 (13.803) | 164.00 (NA) — One participant | 180.30 (NA) — One participant |  |  |  | 173.73 (12.125)
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 49 | 12 | 94
    Phase 2 |  |  |  |  |  |  |  |  |  | 170.98 (8.724) | 169.23 (8.847) | 172.02 (4.183) | 170.14 (8.323)
Weight [Mean (Standard Deviation); unit: kg] — Population: Three patients in Part 2 were diagnosed incorrectly resulting in assignment to the incorrect cohort. These patients are not included in the cohort summaries.
  kg
    Phase 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 0 | 0 | 0 | 22
    Phase 1 | 84.10 (NA) — One participant | 84.10 (NA) — One participant | 72.70 (NA) — One participant | 104.70 (NA) — One participant | 120.10 (NA) — One participant | 72.93 (15.336) | 72.45 (13.307) | 62.90 (NA) — One participant | 110.70 (NA) — One participant |  |  |  | 78.65 (18.333)
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 49 | 12 | 94
    Phase 2 |  |  |  |  |  |  |  |  |  | 70.47 (17.877) | 73.57 (16.527) | 83.83 (13.355) | 74.16 (17.214)

OUTCOME MEASURES:

1. Primary Outcome: Determine the RPII Dose of NC-6004 in Combination With Gemcitabine
Description: In the dose-escalation phase of the study (Part 1), to determine the dose-limiting toxicities (DLTs), MTD, and RPII dose of NC-6004 in combination with gemcitabine
Time Frame: 1 year
Population: Number of participants with at lease one DLT
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 NC-6004 60 mg/m^2 | Phase 1 NC-6004 75 mg/m^2 | Phase 1 NC-6004 90 mg/m^2 | Phase 1 NC-6004 105 mg/m^2 | Phase 1 NC-6004 120 mg/m^2 | Phase 1 NC-6004 135 mg/m^2 | Phase 1 NC-6004 150 mg/m^2 | Phase 1 NC-6004 165 mg/m^2 | Phase 1 NC-6004 180 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1

2. Primary Outcome: Activity of NC-6004 Measured by Progression-free Survival (PFS)
Description: In the expansion phase of the study (Part 2), to evaluate the activity of NC-6004 in combination with gemcitabine in patients with first-line Stage IV squamous NSCLC, first-line advanced or metastatic biliary tract cancer, and first-line metastatic or locally advanced bladder cancer compared with historical control as measured by local investigator/radiologist-assessed progression-free survival (PFS), according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Phase 2 Cohort 1 (NSCLC): Participants with non-small-cell lung cancer (NSCLC) received intravenous (IV) infusion of NC-6004 135 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles for up to 6 cycles.
Arm/Group | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Number analyzed (Participants) | 34 | 50 | 13
days | 116.0 [84.0 to 182.0] | 128.0 [86.0 to 181.0] | 204.0 [130.0 to 233.0]

3. Secondary Outcome: ORR
Description: To evaluate ORR, DCR (DCR = complete response [CR] + partial response [PR] + stable disease [SD]), DOR, PFS, and OS
Time Frame: Up to 40 weeks
Population: This outcome measure was conducted for Phase 2 Arms only as per the Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Number analyzed (Participants) | 34 | 50 | 13
Participants | 4 | 4 | 3

4. Secondary Outcome: DCR
Description: To evaluate ORR, DCR (DCR = complete response [CR] + partial response [PR] + stable disease [SD]), DOR, PFS, and OS
Time Frame: Up to 40 weeks
Population: This outcome measure was conducted for Phase 2 Arms only as per the Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Number analyzed (Participants) | 34 | 50 | 13
Participants | 12 | 19 | 7

5. Secondary Outcome: DOR
Description: To evaluate ORR, DCR (DCR = complete response [CR] + partial response [PR] + stable disease [SD]), DOR, PFS, and OS
Time Frame: every 6 weeks tumor assessments for response and disease progression after treatment discontinuation and telephone calls for survival every 12 weeks until disease progression.
Population: This outcome measure was conducted for Phase 2 Arms only as per the Statistical Analysis Plan.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Number analyzed (Participants) | 4 | 4 | 3
days | 232.0 [227.0 to 281.0] | NA [NA to NA] — Median duration of response and 95% confidence interval was not able to be determined due to an insufficient number of participants with events. | 133.0 [131.0 to 165.0]

6. Secondary Outcome: OS
Description: To evaluate ORR, DCR (DCR = complete response [CR] + partial response [PR] + stable disease [SD]), DOR, PFS, and OS
Time Frame: as for outcome 5
Population: This outcome measure was conducted for Phase 2 Arms only as per the Statistical Analysis Plan.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Number analyzed (Participants) | 34 | 50 | 13
days | 275.0 [119.0 to 366.0] | 350.0 [262.0 to 497.0] | 316.0 [196.0 to NA] — Upper limit of 95% confidence interval was not able to be determined due to an insufficient number of participants with events.

7. Secondary Outcome: EORTC QLQ-C30
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) has the 5 functional scales (physical, role, emotional, cognitive, social), and 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). All of the scales and single item measures range in score from 0 to 100. A positive value of change from baseline means a better outcome in functional scales and a worse outcome in symptom scales.
Time Frame: 1 year
Population: This outcome measure was conducted for Phase 2 Arms only as per the Statistical Analysis Plan.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phase 2 Cohort 2 (Biliary Tract Cancer): Participants with biliary tract cancer received intravenous (IV) infusion of NC-6004 135 mg/m^2 on Day 1 and gemcitabine 1250 mg/m^2 on Days 1 and 8 in 3-week treatment cycles for up to 8 cycles.
Arm/Group | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
Number analyzed (Participants) | 34 | 50 | 13
score on a scale
  Physical Functioning Scale: number analyzed (Participants) | 23 | 40 | 12
  Physical Functioning Scale | -16.522 (20.8767) | -14.000 (18.7835) | -12.222 (22.3531)
  Role Functioning Scale: number analyzed (Participants) | 23 | 40 | 12
  Role Functioning Scale | -10.870 (27.3440) | -13.750 (33.7342) | -18.056 (21.8562)
  Emotional Functioning Scale: number analyzed (Participants) | 23 | 40 | 12
  Emotional Functioning Scale | -2.536 (22.3938) | -1.667 (22.8958) | -10.648 (32.0641)
  Cognitive Functioning Scale: number analyzed (Participants) | 23 | 40 | 12
  Cognitive Functioning Scale | -5.797 (19.2069) | -0.833 (20.9972) | 2.778 (24.4467)
  Social Functioning Scale: number analyzed (Participants) | 23 | 40 | 12
  Social Functioning Scale | -7.971 (32.9024) | -13.333 (30.9397) | -5.556 (21.7113)
  Fatigue: number analyzed (Participants) | 23 | 40 | 12
  Fatigue | 11.594 (17.5613) | 14.444 (28.4895) | 13.889 (28.0792)
  Nausea/Vomiting: number analyzed (Participants) | 23 | 40 | 12
  Nausea/Vomiting | 10.870 (13.8614) | 10.417 (25.2304) | -4.167 (10.3597)
  Pain: number analyzed (Participants) | 23 | 40 | 12
  Pain | 8.696 (26.5288) | 5.833 (30.5575) | 6.944 (20.6685)
  Dyspnoea: number analyzed (Participants) | 23 | 40 | 12
  Dyspnoea | 4.348 (23.1472) | 6.667 (28.4450) | 0.000 (28.4268)
  Insomnia: number analyzed (Participants) | 23 | 40 | 12
  Insomnia | -1.449 (27.4842) | 12.500 (29.8977) | 11.111 (25.9500)
  Appetite Loss: number analyzed (Participants) | 23 | 40 | 12
  Appetite Loss | 15.942 (29.9319) | 9.167 (43.3547) | 2.778 (17.1643)
  Diarrhoea: number analyzed (Participants) | 23 | 40 | 12
  Diarrhoea | 5.797 (12.9184) | 0.833 (14.0967) | 0.000 (0.0000)
  Financial Difficulties: number analyzed (Participants) | 23 | 40 | 12
  Financial Difficulties | 10.145 (21.1650) | 5.833 (22.5036) | 2.778 (17.1643)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Phase 1 NC-6004 60 mg/m^2 | Phase 1 NC-6004 75 mg/m^2 | Phase 1 NC-6004 90 mg/m^2 | Phase 1 NC-6004 105 mg/m^2 | Phase 1 NC-6004 120 mg/m^2 | Phase 1 NC-6004 135 mg/m^2 | Phase 1 NC-6004 150 mg/m^2 | Phase 1 NC-6004 165 mg/m^2 | Phase 1 NC-6004 180 mg/m^2 | Phase 2 Cohort 1 (NSCLC) | Phase 2 Cohort 2 (Biliary Tract Cancer) | Phase 2 Cohort 3 (Bladder Cancer)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 1/9 | 0/6 | 0/1 | 0/1 | 21/34 | 30/50 | 9/13
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 4/9 | 3/6 | 1/1 | 1/1 | 13/34 | 17/50 | 4/13
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 9/9 | 6/6 | 1/1 | 1/1 | 34/34 | 50/50 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 NC-6004 60 mg/m^2 (N=1) | Phase 1 NC-6004 75 mg/m^2 (N=1) | Phase 1 NC-6004 90 mg/m^2 (N=1) | Phase 1 NC-6004 105 mg/m^2 (N=1) | Phase 1 NC-6004 120 mg/m^2 (N=1) | Phase 1 NC-6004 135 mg/m^2 (N=9) | Phase 1 NC-6004 150 mg/m^2 (N=6) | Phase 1 NC-6004 165 mg/m^2 (N=1) | Phase 1 NC-6004 180 mg/m^2 (N=1) | Phase 2 Cohort 1 (NSCLC) (N=34) | Phase 2 Cohort 2 (Biliary Tract Cancer) (N=50) | Phase 2 Cohort 3 (Bladder Cancer) (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 NC-6004 60 mg/m^2 (N=1) | Phase 1 NC-6004 75 mg/m^2 (N=1) | Phase 1 NC-6004 90 mg/m^2 (N=1) | Phase 1 NC-6004 105 mg/m^2 (N=1) | Phase 1 NC-6004 120 mg/m^2 (N=1) | Phase 1 NC-6004 135 mg/m^2 (N=9) | Phase 1 NC-6004 150 mg/m^2 (N=6) | Phase 1 NC-6004 165 mg/m^2 (N=1) | Phase 1 NC-6004 180 mg/m^2 (N=1) | Phase 2 Cohort 1 (NSCLC) (N=34) | Phase 2 Cohort 2 (Biliary Tract Cancer) (N=50) | Phase 2 Cohort 3 (Bladder Cancer) (N=13)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 4 | 4 | 1 | 1 | 6 | 15 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 6 | 6 | 1 | 1 | 5 | 15 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 1 | 1 | 0 | 7 | 1
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 1 | 1 | 7 | 12 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 4 | 3 | 1 | 1 | 0 | 15 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 5 | 2 | 1 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 1 | 4 | 3 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 6 | 3 | 0 | 1 | 1 | 8 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 3 | 2
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 0 | 0 | 6 | 4 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 1 | 1 | 7 | 14 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 4 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 5 | 5 | 1 | 0 | 5 | 8 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1 | 9 | 6 | 1 | 1 | 17 | 24 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 5 | 3 | 1 | 1 | 7 | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 1 | 4 | 13 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 2 | 1 | 0 | 2 | 7 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 9 | 4 | 1 | 1 | 16 | 32 | 8
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 1 | 0 | 7 | 24 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 6 | 6 | 1 | 1 | 16 | 18 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 3 | 3 | 1 | 0 | 11 | 11 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 5 | 13 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 6 | 3 | 1 | 1 | 3 | 16 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 4 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 8 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 5 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 8 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 5 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT02240238/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT02240238/SAP_001.pdf